CLINICAL TRIAL: NCT00450931
Title: Helping Patients and Physicians Make Sense of Medical Data
Brief Title: Drug Facts Page or a Short Drug Summary in Helping Patients and Doctors Understand Medical Information
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: White River Junction Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized
Other Study IDs: CDR0000513888; VAMC-WRJ-15879; DMS-15879; NCT00386932 (obsolete NCT alias)
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2008-09

CONDITIONS: Health Status Unknown
Keywords: health status unknown
MeSH Terms: interventions — Counseling; Early Intervention, Educational

INTERVENTIONS:
Other: counseling intervention
Other: educational intervention

SUMMARY:
RATIONALE: The way in which information about a drug is provided may affect the ability of patients and doctors to understand how a drug works and the side effects of the drug.

PURPOSE: This randomized trial is studying how well a drug facts page works compared with a standard brief summary in helping patients and doctors understand medical information.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the effect of a prescription drug summary (one-page summary of drug information that includes a table with data on drug benefit and side effects) vs standard brief summary in direct-to-consumer advertisements on the comparisons of two drugs for the same indication, knowledge of drug efficacy and side effects of each drug.

Secondary

* Comprehension of information contained in the drug facts box and rating of the usability of the drug information.

OUTLINE: This is a randomized study. Participants are contacted by phone via random-digit dialing for initial interview using the computer-assisted telephone interviewing (CATI) system. Eligible participants are then randomized to 1 of 4 intervention arms.

* Arm I: Participants receive 2 advertisements for a drug to treat heartburn with a drug facts second page.
* Arm II: Participants receive 2 advertisements as in arm I for drugs to treat heatburn with the standard second page (i.e., brief summary).

Participants in both arms complete the self-reported questionnaire mailed with the advertisement intervention.

PROJECTED ACCRUAL: A total of 200 participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* English-speaking adults
* Must be able to be chosen by Random Digit Dialing

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)

PRIMARY OUTCOMES:
Comparison of two drugs for the same indication
Knowledge of drug efficacy and side effects of each drug

SECONDARY OUTCOMES:
Comprehension of information contained in the drug facts box and rating of the usability of the drug information

CONTACTS AND LOCATIONS:
Overall Officials: Steven Woloshin, MD, MS, Principal Investigator — White River Junction Veterans Affairs Medical Center; Harold Bae — White River Junction Veterans Affairs Medical Center